CLINICAL TRIAL: NCT01874470
Title: Renal Denervation by Allegro System in Patients With Resistant Hypertension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai AngioCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Allegro-HTN
Record Dates: First submitted 2013-06-01; First posted 2013-06-11 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2013-12

CONDITIONS: Renal Denervation; Resistant Hypertension; Standard Medication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard medication (Placebo Comparator): Standard Medication: Continued usage of 3 or more antihypertensive medications of different classes, including a diuretic
  Interventions: Other: standard medication
- renal denervation (Experimental): Allegro Renal Denervation System (AngioCare)
  Interventions: Device: renal denervation; Other: standard medication

INTERVENTIONS:
Device: renal denervation
  Other Names: Allegro Renal Denervation System (AngioCare)
  Arms: renal denervation
Other: standard medication
  Other Names: Standard Medication: Continued usage of 3 or more antihypertensive medications of different classes, including a diuretic

SUMMARY:
The purpose of ALLEGRO-HTN trial is to evaluate the safety and effectiveness of renal denervation in subjects with resistant hypertension by using Allegro renal denervation system

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years at time of randomization
* Stable medication regimen including 3 or more antihypertensive medications of different classes, including a diuretic (with no changes for a minimum of 4 weeks prior to screening) and no expected changes for at least 6 months
* 1) Office SBP and/or DBP ≥160/100 mm Hg ( ≥ 150/95 mmHg for type II diabetic patients) , 2) ABPM 24 hour average SBP and/or DBP ≥140 and/or 90 mmHg
* Main renal arteries with ≥4 mm diameter or with ≥20 mm treatable length (by visual estimation)
* eGFR≥45 mL/min/1.73 m2
* Written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* Secondary hypertension
* Has an implantable cardioverter defibrillator (ICD) or pacemaker
* Myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within 6 months of the screening period
* Intravascular thrombosis or unstable atherosclerotic plaques
* Has hemodynamically significant valvular heart disease
* Pregnant, nursing, or planning to be pregnant
* Any serious medical condition that may adversely affect the safety of the participant or the study
* Currently enrolled in another investigational drug or device trial

Angiographic Exclusion Criteria:

* Renal artery stenosis (≥50%) or renal artery aneurysm in either renal artery
* History of prior renal artery intervention including balloon angioplasty or stenting
* Multiple renal arteries where the main renal artery is estimated to supply <75% of the kidney
* Main renal arteries with <4 mm diameter or with <20 mm treatable length (by visual estimation)
* Renal artery abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in office-based systolic blood pressure (SBP) from baseline to 6 months | 6 month

SECONDARY OUTCOMES:
Change in average 24-hour SBP by ambulatory blood pressure monitoring (ABPM) from baseline to 6 months | 6 month
  Change in average 24-hour SBP by ambulatory blood pressure monitoring (ABPM) from baseline to 6 months
• The incidence of major adverse events (MAE) at 1 month postrandomization | 1-month post randomization
Office SBP and DBP at 1, 3, 6 months postrandomization | up to 6 months
• Patient-recorded home systolic blood pressure at 1, 3, 6 months postrandomization | up to 6 months
• MAE at 6-month post-randomization, including new renal artery stenosis >60% | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, China